CLINICAL TRIAL: NCT00430534
Title: To Evaluate the Safety, Immunogenicity and Efficacy of GSK Biologicals' EBV Vaccine (268664) in Healthy Seronegative Adolescents/Adults When Injected Intramuscularly According to a 0-1-5 Month Schedule in Belgium.
Brief Title: Evaluation of Safety, Immune-Response and Efficacy of GSK Biologicals' EBV (Epstein Barr Virus) Vaccine (268664).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Henogen (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HN/P001-EBV-003
Record Dates: First submitted 2007-02-01; First posted 2007-02-02 (Estimated); Last update posted 2007-02-02 (Estimated); Status verified 2007-02

CONDITIONS: Epstein Barr Virus (EBV) Infection
Keywords: Epstein Barr Virus; Belgium; Infectious mononucleosis
MeSH Terms: conditions — Epstein-Barr Virus Infections; Infections; Infectious Mononucleosis

INTERVENTIONS:
Biological: EBV vaccine (268664)

SUMMARY:
To evaluate the safety, immune-response and efficacy of GSK Biologicals' EBV vaccine in a population at risk of developing infectious mononucleosis. Each subject will receive three doses of vaccine or placebo during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adolescent/adult subjects between and including 16 and 25 years of age at the time of screening.

  * Written informed consent obtained from the subject prior to enrolment.
  * Seronegative for EBV antibody.

Exclusion Criteria:

* Administration of immunoglobulin and/or any blood products within the three months (90 days) preceding the first dose of study vaccine or planned administration during the study period.

  * Use of any investigational or non-registered drug or vaccine other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
  * Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
  * Family history of congenital or hereditary immunodeficiency.
  * Major congenital defects or serious chronic illness.
  * History of any neurologic disorders or seizures, with the exception of a single febrile seizure during childhood.
  * Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
  * History of intravenous drug abuse within the past 2 years.
  * Known or suspected allergy to any vaccine component.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200

PRIMARY OUTCOMES:
Attack rates of infectious mononucleosis over 18 months after Dose 2

SECONDARY OUTCOMES:
Solicited symptoms (Day 0-7); unsolicited AEs (Day 0-29 ); SAEs (full study)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Henogen
Locations (1):
- GSK Clinical Trials Call Center, Brussels, Belgium

REFERENCES:
- [Derived] Sokal EM, Hoppenbrouwers K, Vandermeulen C, Moutschen M, Leonard P, Moreels A, Haumont M, Bollen A, Smets F, Denis M. Recombinant gp350 vaccine for infectious mononucleosis: a phase 2, randomized, double-blind, placebo-controlled trial to evaluate the safety, immunogenicity, and efficacy of an Epstein-Barr virus vaccine in healthy young adults. J Infect Dis. 2007 Dec 15;196(12):1749-53. doi: 10.1086/523813. PMID 18190254